CLINICAL TRIAL: NCT06602388
Title: Non-interventional, Monocentric Study Aimed at Building up a Collection of Biological Samples Collected From Bioaster Collaborators for Scientific Purposes
Brief Title: Human Internal BIOASTER's Samples Collection
Acronym: HIBISCUS
Status: Not yet recruiting | Type: Observational
Sponsor: Bioaster (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-A00323-44
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Biological Samples
Keywords: Biological; samples; collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — biological samples: stool, urine, saliva, buccal swab, nasal swab, superficial skin swab, hair
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy volunteers (Bioaster employees): Collection of biological samples from healthy volunteers: Stool, urine, saliva, buccal swab, nasal swab, superficial skin swab, hair
  Interventions: Other: Biological sampling

INTERVENTIONS:
Other: Biological sampling — Collection of biological samples from healthy volunteers: Stool, urine, saliva, buccal swab, nasal swab, superficial skin swab, hair

SUMMARY:
BIOASTER is a Technological Research Institute dedicated to microbiology and infectious diseases. BIAOSTER s areas of expertise are organized around four research programs: 1/ Antimicrobials; 2/ Vaccines; 3/ Microbiota; 4/ Diagnostics.

Hibiscus is a non-interventional, monocentric study aimed at building up a a collection of biological samples (stool, urine, saliva, buccal swab, nasal swab, superficial skin swab, hair) collected from BIOASTER employees. These samples to be used for scientific purposes including the technological development of Bioaster s collaborative and in-house research projects.

ELIGIBILITY:
Inclusion Criteria:

Some inclusion criteria can be defined according to the needs of the scientific objective. For example, it is up to volunteers to decide whether or not to participate if they meet the following criteria:

* Age criteria (e.g.: specific, non-identifying range sought: 30-40 years)
* BMI criteria (for example: BMI between 18.5 and 29 kg/m2)
* Gender criteria (e.g.: women only)

Exclusion Criteria:

Some of the following non-inclusion criteria may be defined according to the needs of the project:

* Minor subject
* Health criteria (e.g. presence or absence illness/infection/vaccination/allergy/anti-infective treatment in the last 3 months prior to the date of sampling)
* Smoker status
* Severe chronic illness (active cancer, HIV, severe renal failure, ongoing severe heart, liver or biliary disorders, arthritis)
* Diagnosed acute or chronic gastrointestinal disease or complication (e.g. celiac disease, gastroesophageal reflux, gastric or duodenal ulcer, Crohn's disease, hemorrhoids, irritable bowel syndrome),

In all cases, it will be requested that volunteers with the following criteria do not participate in the study:

* Pregnant or breast-feeding women
* Subjects under curatorship or guardianship
* Subjects under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers (Bioaster employees)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of analyzable samples collected for scientific purposes. | 3 years after the first inclusion
  The number of analyzable samples collected for scientific purposes at the end of inclusion periode

CONTACTS AND LOCATIONS:
Overall Officials: Cyril GUYARD, Study Director, Study Director — Bioaster; Dr Xavier MORGE, Principal Investigator — Bioaster

IPD SHARING:
Plan to Share IPD: No